CLINICAL TRIAL: NCT05629377
Title: Hypothalamic Amenorrhea as a Fertility Status Marker for Cardiovascular Health
Brief Title: Hypothalamic Amenorrhea as a Fertility Status Marker for Cardiovascular Health (ARCH)
Acronym: ARCH
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chrisandra L. Shufelt, MD, Principal Investigator, Mayo Clinic
Other Study IDs: 22-006348; R01HD106096 (NIH)
Record Dates: First submitted 2022-10-14; First posted 2022-11-29 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Hypothalamic Amenorrhea
Keywords: Functional Hypothalamic Amenorrhea; Amenorrhea
MeSH Terms: conditions — Amenorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypothalamic amenorrhea (HA) occurs during reproductive years and results in stopped menstrual cycles and infertility which can be prolonged from months to years and is characterized by varying combinations of psychosocial stress, anxiety, high levels of physical activity, and/or weight loss. Data from our group indicates that one-third of women with HA (mean age: 27 yrs) have preclinical cardiovascular disease (CVD) measured noninvasively as vascular dysfunction and vascular inflammation. This study will use HA as a marker of fertility status for cardiovascular health and perform dense-phenotyping using remote patient monitoring (FitBit) and patient reported outcomes (questionnaires) to determine which HA phenotypes are related to preclinical CVD and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Secondary amenorrhea of 3 or more consecutive months duration
* Include the screening hormones (eg, estradiol (E2) < 50 pg/ml, Follicle-Stimulating Hormone (FSH) <10 mIU/ml, and Luteinizing Hormone (LH) < 10mIU/ml and other HA-defining hormones); or clinical diagnosis of HA by medical providers.
* Pre-menopause status.
* Able to give informed consent.

Exclusion Criteria:

* A diagnosis for secondary amenorrhea including prolactinoma, Polycystic Ovary Syndrome (PCOS), premature ovarian insufficiency, pituitary surgery, infection or infarction
* Pregnancy
* Psychotropic/illicit drug use
* Mental/neurological/major psychological disorders (other than depression and anxiety).
* Parturition/lactating in the last 6-12 months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Premenopausal women with hypothalamic amenorrhea at Mayo Clinic Florida.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Hypothalamic Amenorrhea (HA) duration | 3 months
  Duration of HA by month of amenorrhea (absence of menstruation)
Vascular dysfunction | 3 months
  Measured by reactive hyperemic index (RHI)
Psychosocial stress | 3 months
  Measured by NIH PROMIS® short-form questionnaires
Perceived stress | 3 months
  Measured by the validate perceived stress scale questionnaire, a 10-item questionnaire, scores range from 0 to 40; higher scores indicate higher levels of perceived stress.
Step count | 3 months
  Measured by Fitbit Versa 2 watch that tracks steps per day, active and resting heart rate, sleep hours per day
Physical activity level | 3 months
  Measured by Fitbit Versa 2 watch that tracks amount of light physical activity, moderate, and vigorous activity
Heart Rate | 3 months
  Measured by Fitbit Versa 2 watch that tracks heart rate
Caloric intake and nutrition | 3 days
  Measured using a self-reported food diary
Vascular inflammation | 3 months
  concentration of cytokines multiplex immunoassay platform

CONTACTS AND LOCATIONS:
Overall Officials: Chrisandra Shufelt, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20538611